CLINICAL TRIAL: NCT03882346
Title: A Phase 2b Study to Evaluate Safety and Efficacy of LifeLiver (Bio Artificial Liver) in Acute or Acute-on-Chronic Liver Failure Patients Waiting Emergent Liver Transplantation
Brief Title: Study to Evaluate Safety and Efficacy of LifeLiver in Acute or Acute-on-Chronic Liver Failure Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HLB Cell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC-BAL-18
Record Dates: First submitted 2019-03-13; First posted 2019-03-20 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Acute Liver Failure; Acute-On-Chronic Liver Failure
Keywords: Acute Liver Failure; Acute-On-Chronic Liver Failure; Artificial Liver; Liver Transplantation
MeSH Terms: conditions — Liver Failure, Acute; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Intervention Model Description: This is a parallel, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in Control Group will receive best supportive care for the disease.
- Experimental Group (Experimental): Patients in Experimental Group will receive LifeLiver treatment in addition to best supportive care for the disease.
  Interventions: Combination Product: LifeLiver

INTERVENTIONS:
Combination Product: LifeLiver — LifeLiver is an extracorporeal bioartificial liver (BAL) system. The system has shown remarkable detoxification capacity and sustained hepatic functions and also provides a bridge to transplant for patients who are unable to receive timely liver transplantation.
  Arms: Experimental Group

SUMMARY:
This is a prospective, comparative, open label, phase 2b study designed to investigate the safety and efficacy of LifeLiver (an Extracorporeal Bio Artificial Liver). The study will recruit approximately 40 acute or acute-on-chronic liver failure patients.

DETAILED DESCRIPTION:
Patient should have acute or acute-on-chronic liver failure and be registered in KONOS (Korean Network for Organ Sharing) system as a candidate of liver transplantation. Patients who meet the eligibility criteria will be assigned to control group or experimental group. Experimental group patients will receive LifeLiver treatment in addition to the best supportive care for the disease.

Primary Objective:

1. To evaluate the efficacy of LifeLiver in terms of a comparison of 30 day-survival rate between control group and experimental group. (after patient's KONOS (Korean Network for Organ Sharing) registration date)

Secondary Objective:

1. To compare a median value of 2 week-survival rate and duration of survival between both study groups
2. Survival analysis respect to each group of patients divided according to the KONOS status
3. To investigate safety and change of overall efficacy indicators in terms of Glasgow Coma Scale, West Heaven Criteria for hepatic encephalopathy, MELD (Model for End-stage Liver Disease) score, blood ammonia, inflammatory cytokine

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age
* Acute or acute-on-chronic liver failure patients who is waiting for liver transplantation (KONOS liver transplant emergency grade 2 or 3)
* Hepatic encephalopathy grade II or above
* The following laboratory values must be documented within the screening period:

  * INR (international normalized ratio) 2.0 or above
  * Serum ammonia 56 micromole/L or above
  * Total bilirubin 5mg/dL or above
  * Body weight 45kg or above
* Patient who can not expect effective treatment or prolonged survival
* Patient or patient's legal representative willing to provide informed consent and commit to study procedures

Exclusion Criteria:

* Patient who has contraindication to plasmapheresis
* Severe hypotension (systolic blood pressure 80mmHg or less)
* Platelet < 15,000/mm3
* Contraindications to liver transplantation (sepsis, severe heart disease, uncontrollable hemorrhage, irreversible brain damage)
* Cerebral hemorrhage
* Positive HIV infection
* Serious or life-threatening hemorrhage just before initiation of the study
* Patients with high gastrointestinal bleeding tendency (a history or suspicion of gastrointestinal bleeding within last 3 months)
* Hepatocellular carcinoma patient with 7 (or more) tumors or a 6cm (or larger) diameter single tumor
* Pregnant or lactating women
* Antibiotics (beta-lactam family) hypersensitive and streptomycin, amphotericin B sensitive patients
* Patients with inappropriate condition to participate the study under investigator's judgement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Survival rate for 30 days | up to 30 days
  To compare survival rate of LifeLiver treatment with best supportive care
Occurrence of clinical safety laboratory adverse events (AEs) | up to approximately 12 months
  To compare occurrence of clinical safety laboratory adverse events between Experimental group and Control group assessed according to NCI-CTCAE v5.0
Incidence of transition of PERV (Porcine Endogenous Retrovirus) (for experimental group only) | up to approximately 12 months
  Number of reported PERV transition defined as viral detection in subject's blood by PCR (Polymerase Chain Reaction) test.

SECONDARY OUTCOMES:
Survival rate for 14 days | up to 14 days
  To compare survival rate of LiveLiver treatment with best supportive care
Median value of duration of survival | up to approximately 12 months
  To compare Median value of duration of survival between experimental group and control group
Kaplan-Meier estimate of subjects with MELD (Modell for End-stage Liver Disease) score >37 | up to 30 days
  To compare Kaplan-Meier estimate of both (experimental and control) groups at 14 days and 30 days
Kaplan-Meier estimate of subjects with 31≤ MELD score ≤37 | up to 30 days
  To compare Kaplan-Meier estimate of both groups at 14 days and 30 days
Comparison of MELD score | up to approximately 12hours after completion of LifeLiver treatment
  Intra-group comparison (between pre and post 12 hours of LifeLiver treatment) and Inter-group comparison (between both groups) of subject's MELD score (range of minimum 6 to maximum 40)
Comparison of subject's neurological status - hepatic encephalopathy grade | up to approximately 12 hours after completion of LifeLiver treatment
  Intra-group comparison (between pre and post 12 hours of LifeLiver treatment) and Inter-group comparison (between both groups) of subject's hepatic encephalopathy grade (range of minimum 1 to maximum 4)
Comparison of subject's neurological status - Glasgow Coma Scale | up to approximately 12 hours after completion of LifeLiver treatment
  Intra-group comparison (between pre and post 12 hours of LifeLiver treatment) and Inter-group comparison (between both groups) of subject's Glasgow Coma Scale (range of minimum 3 to maximum 15)
Comparison of subject's value of blood ammonia | up to approximately 12 hours after completion of LifeLiver treatment
  Intra-group comparison (between pre and post 12 hours of LifeLiver treatment) and Inter-group comparison (between both groups) of subject's value of blood ammonia
Comparison of subject's value of inflammatory cytokines | up to approximately 12 hours after completion of LifeLiver treatment
  Intra-group comparison (between pre and post 12 hours of LifeLiver treatment) and Inter-group comparison (between both groups) of subject's value of inflammatory cytokines (TNF-α, Interleukin-6, Interleukin-10)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hyun Sinn, MD, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea